CLINICAL TRIAL: NCT05575505
Title: Phosphodiesterase Inhibitors, Pentoxifylline, as Adjunctive Therapy in Patients With Ulcerative Colitis.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/2022
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Mesalamine group, who will receive 1 g mesalamine three times daily for 6 months.
- Pentoxifylline group (Active Comparator): The pentoxifylline group will receive 1 g mesalamine three times daily plus pentoxifylline 400 mg two times daily for 6 months.
  Interventions: Drug: Pentoxifylline 400 MG

INTERVENTIONS:
Drug: Pentoxifylline 400 MG — Pentoxifylline (PTX) is a methyl-xanthine derivative that possesses antioxidant and anti-inflammatory characteristics
  Arms: Pentoxifylline group

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease characterized by diffused inflammation of the colon and rectum mucosa; however, the exact underlying mechanisms of UC remain poorly understood. Also, it is associated with high risk of colon cancer, so there is a continuous need for introducing new therapies that decrease progression, and hence better outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both males and females will be included
* Negative pregnancy test and effective contraception.

Exclusion Criteria:

* Breastfeeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies
* Addiction to alcohol and / or drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
changes in Mayo Score Index. | 6 months
  The Mayo Score for ulcerative colitis disease activity assesses disease severity and can be used to monitor patients during therapy.
  This scale uses four parameters to calculate the patient scores from 0-12. The parameters assessed are rectal bleeding, stool frequency, endoscopic findings, and physician assessment. Higher scores mean poor progression. Lower scores mean good progression

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt